CLINICAL TRIAL: NCT07155967
Title: Effect of Cross-Education in Blood Flow Restriction Resistance Training on Lower Limbs in Older Women: A Randomized Controlled Clinical Trial
Brief Title: Effect of Cross-Education in Blood Flow Restriction Resistance Training on Lower Limbs in Older Women
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Franciele Marques Vanderle, Principal Investigator, Paulista University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 86845325.1.0000.5402
Record Dates: First submitted 2025-08-14; First posted 2025-09-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Muscle Strength; Hypertrophy
Keywords: Elderly population; Strength training; Physical exercise; Lower limb; Blood flow restriction therapy
MeSH Terms: conditions — Hypertrophy; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-intensity unilateral resistance training group with blood flow restriction (Experimental): This group will perform the training protocol, with the dominant lower limb (LL) executing the exercises using an occlusion cuff set at 40% of total occlusion pressure (TOP), applied continuously throughout the session, while the other limb will perform the exercises without BFR.
  Interventions: Device: Blood Flow Restriction Cuff
- Low-intensity bilateral resistance training group without blood flow restriction (No Intervention): This group will perform the training protocol on both limbs (bilaterally) without the use of blood flow restriction (BFR).

INTERVENTIONS:
Device: Blood Flow Restriction Cuff — Inflatable device that exerts an external pressure above a muscle or joint of the extremities.
  Arms: Low-intensity unilateral resistance training group with blood flow restriction

SUMMARY:
Unilateral resistance training has been shown to promote strength adaptations in the directly trained limb and also improve strength in the contralateral limb, a phenomenon known as cross-education (CE), with more pronounced effects observed in high-load training. However, high-load resistance training may be unfeasible for older adults. Blood flow restriction (BFR) training emerges as a low-load alternative that reduces joint stress, is easy to apply, and has low cost. Although there is already evidence showing significant effects of CE during resistance training with BFR, gaps remain regarding its applicability in older adults. This study aims to evaluate the effects of CE in resistance training with BFR on the lower limbs of older women.

DETAILED DESCRIPTION:
A randomized controlled clinical trial will be conducted with 32 older women aged 60 years or older. Participants will be randomly assigned to one of two groups: a low-intensity unilateral resistance training group with blood flow restriction (BFR) (experimental group) and a low-intensity unilateral resistance training group without BFR (control group). Baseline assessments will include the following: pain using the Visual Analog Scale (VAS); perception of recovery and discomfort using the Likert scale; perceived exertion using the Borg CR-10 scale; systolic and diastolic blood pressure measured via the auscultatory method; heart rate using a Polar portable heart rate monitor; oxygen saturation via pulse oximetry; quadriceps circumference using a measuring tape; muscle mass assessed by ultrasound; muscle tone, stiffness, and elasticity evaluated by myotonometry; cellular health and integrity using bioelectrical impedance analysis (BIA); functional performance through the Timed Up and Go test (TUG), the Short Physical Performance Battery (SPPB), and a test of agility and dynamic balance (AGIL); and muscle strength measured by the one-repetition maximum test (1RM). Following the baseline assessment, participants will undergo the training protocol according to their group assignment. Hemodynamic parameters-heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), and oxygen saturation (SpO₂)-as well as perceptual measures (VAS, Likert scale, and CR-10) will be collected before and immediately after each training session. After three weeks of training, an intermediate evaluation of all outcomes will be performed, along with load adjustment. Following this, participants will complete an additional three weeks of training. One week after the conclusion of the intervention, a final evaluation of all outcomes will be conducted. Descriptive statistics and repeated-measures ANOVA will be used for data analysis, with a significance level set at p < 0.05.

Participants will be duly informed about the procedures and objectives of this study, and after agreeing, they will sign an informed consent form, effectively becoming part of it. In the consent form, participants will be asked if they agree to the use of their data if they choose to withdraw from the study. Participants will also be asked for permission for the research team to share relevant data with people at universities participating in the research or regulatory authorities, where relevant. The study were approved to the Research Ethics Committee of FCT/UNESP, Presidente Prudente, SP, Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Elderly women who present one or more of the following characteristics will not be included:

  1. a history of stroke, progressive neurological disease, or dementia;
  2. communication difficulties due to aphasia or hearing loss;
  3. any health condition that contraindicates or prevents physical exercise;
  4. a history of hip or knee surgery (e.g., arthroscopy or arthroplasty) or recent lower limb musculoskeletal injury that could impair performance during tests or training (e.g., osteoarthritis, osteoporotic fracture, muscle injury, and/or back pain in the past six months);
  5. use of supplements aimed at improving physical performance and/or muscle mass; or
  6. one or more predisposing risk factors for thromboembolism.

Exclusion Criteria:

Participants will be excluded from the study if they use medications (analgesics or anti-inflammatory drugs) or other therapeutic interventions that could interfere with any outcomes, or if they sustain an injury resulting from the training and choose to withdraw from the study.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals assigned female at birth will be included, due to physiological characteristics relevant to the study objectives.
Enrollment: 32 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Muscle strength assessment | 3 days (baseline, mid-intervention, and final assessment)
  The one-repetition maximum (1RM) test will be used to assess muscle strength, as well as to prescribe the training protocol. It will be performed bilaterally during the initial, intermediate, and final assessments. Initially, participants will perform one repetition to familiarize themselves with the knee extension movement, followed by 10 warm-up repetitions using a load of 30-40% of the estimated 1RM. After the warm-up, the test will begin with a load equivalent to 20% of the participant's body mass, considering the target muscle group (quadriceps muscle). Load will then be progressively increased by 5-10% with each attempt. The participant must perform only one repetition per attempt. If successful, a rest interval of 3 to 5 minutes will be given before the next load increment and attempt. The 1RM is defined as the highest load the participant can lift once with proper form, without any compensatory movements. The test is considered valid if the participant reaches their maximum.
Ultrasound | 3 days (baseline, mid-intervention, and final assessment)
  The assessment of the muscular structure will be carried out using ultrasound images of the participant's lower limbs, which will be captured using BodyMetrix BX-2000. Participants will be assessed in the supine position with legs fully extended and muscles relaxed. The ultrasound transducer will be covered with water-soluble transmission gel and positioned perpendicular to the skin over the muscle.
Quadriceps circumference | 3 days (baseline, mid-intervention, and final assessment)
  Thigh circumference measurements will be taken at the proximal, medial, and distal positions, with the participant standing upright, heels approximately 10 cm apart, and body weight evenly distributed between both feet. For all measurements, the evaluator should position themselves so that their line of sight is level with the measurement site. Three non-consecutive measurements will be performed at each site, and the highest value will be recorded. A marker pen will be used to identify the exact anatomical locations for measurement.
Arterial pressure | 9 weeks (at baseline, mid-intervention, and post-intervention, as well as before and immediately after training sessions)
  It will be collected with a sphygmomanometer
Heart rate | 9 weeks (at baseline, mid-intervention, and post-intervention, as well as before and immediately after training sessions)
  Heart rate will be continuously monitored using a portable heart rate monitor, Polar® RS800cx model (Polar Electro OY, Finland).
Oxygen saturation | 9 weeks (at baseline, mid-intervention, and post-intervention, as well as before and immediately after training sessions)
  Oxygen saturation will be measured using a fingertip pulse oximeter (ChoiceMMED - MD300C1 Fingertip, China), attached to the right index finger of each participant.
Subjective Pain Assessment | 9 weeks (at baseline, mid-intervention, and post-intervention, as well as before and immediately after training sessions)
  Subjective pain assessment will be obtained using the Visual Analog Scale (VAS), graded from 0 to 10, with zero indicating no pain and 10 representing the maximum level of pain tolerated by the participant, as described by Ferreira et al. Participants will be asked about the presence of pain in the dominant and non-dominant lower limbs, identifying on the scale the number corresponding to their current pain intensity.
Subjective Perception of Discomfort | 6 weeks (immediately after the training sessions)
  Subjective perception of discomfort will be assessed using the Borg CR-10 scale, representing the perception of discomfort, with 0 corresponding to "no discomfort" and 10 to "maximum discomfort." Participants will be asked to report the discomfort perceived immediately after unilateral training with blood flow restriction (BFR). It should be noted that although the Borg CR-10 scale is not specifically designed for this purpose, it is commonly used in the BFR literature. The scale will be presented to participants in a way that prevents influence from the researcher.
Subjective Perception of Recovery | 9 weeks (at baseline, mid-intervention, and post-intervention, as well as before and immediately after training sessions)
  Subjective perception of recovery of the lower limb subjected to the exercise protocol will be assessed using a 10-point Likert scale, where 1 indicates "not recovered" and 10 "fully recovered." The scale will be presented to participants in a way that prevents influence from the researcher. The question will first be asked for the dominant lower limb and subsequently for the non-dominant lower limb.
Subjective Perception of Effort | 9 weeks (at baseline, mid-intervention, and post-intervention, as well as before and immediately after training sessions)
  The Borg Rating of Perceived Exertion (RPE) scale (45) is an instrument used to assess the subjective perception of effort generated during a given activity. This instrument, proposed by Borg, consists of a 0 to 10-point scale (CR-10), where participants select the descriptor and number that best reflect their psychophysiological stress related to the exercise. Before the exercise, participants will receive instructions on how to accurately respond to the RPE scale. Participants will report their perceived effort while looking at the scale, where 0 indicates "no effort" and 10 indicates "maximal effort."
Myotonometry | 9 weeks (at baseline, mid-intervention, and post-intervention, as well as before and immediately after training sessions)
  Muscle tone, stiffness, and elasticity of the quadriceps femoris will be assessed using the MyotonPRO® device (MyotonAS, Tallinn, Estonia). The device will be positioned at two-thirds of the distance between the anterior superior iliac spine (ASIS) and the superior pole of the patella, 4 cm above the base of the patella, 15 cm below the ASIS, at the midpoint between the patella and the anterior inferior iliac spine (AIIS), and 2 cm medially and 2 cm laterally from the midpoint. The device will be placed perpendicular to the assessed region, applying a light pre-load pressure, controlled at 0.18 N of initial compression of the subcutaneous tissue. Subsequently, an additional impulse of 0.40 N will be released for 15 ms, inducing tissue oscillation, which will then be dampened or attenuated.
Bioelectrical impedance analysis | 9 weeks (at baseline, mid-intervention, and post-intervention, as well as before and immediately after training sessions)
  Bioimpedance will be measured using a tetrapolar device (BIA Analyzer, 50 kHz, 800 µA). Electrodes will be positioned on the quadriceps femoris muscles. Analyzed variables will include resistance (R), reactance (Xc), phase angle (PhA), and tolerance ellipse, via Bioscan software.
Functional mobility | 3 days (baseline, mid-intervention, and final assessment)
  The Timed Up and Go (TUG) test is a simple and quick physical test used to assess and classify functional mobility and fall risk in older adults. A time of up to 10 seconds is considered normal for healthy and independent individuals; 11 to 20 seconds are considered partially independent, with impairment and/or low risk of falls; 21 to 29 seconds indicates a moderate risk of falls; and more than 30 seconds suggests impaired physical mobility and a high risk of falls.
Physical performance | 3 days (baseline, mid-intervention, and final assessment)
  The Short Physical Performance Battery (SPPB) assesses physical performance and includes three domains: semi-static balance, lower limb strength, and gait speed. Each test has a maximum score of 4 points, and the total score is the sum of the three tests, with a maximum of 12 points. The final classification is as follows: 0-3 points - disability or poor performance; 4-6 points - low performance; 7-9 points - moderate performance; 10-12 points - good performance.
Agility and dynamic balance test | 3 days (baseline, mid-intervention, and final assessment)
  The Agility and Dynamic Balance (AGIL) test is part of the AAHPERD test battery, in which tasks similar to daily functional fitness activities are performed. Reference values for older women: 10.3-19.5 seconds - very good; 19.6-21.4 seconds - good; 21.5-23.6 seconds - fair; 23.7-26.4 seconds - poor; 26.5-44.4 seconds - very poor.

OTHER OUTCOMES:
Occlusion pressures (AOP) | Baseline
  To determine the AOP, the Doppler equipment transducer will be used, which will be positioned over the posterior tibial artery to capture the auscultatory pulse. A blood pressure cuff will be fixed to the participant's thigh close to the region of the inguinal fold of the dominant limb, and then with the inflatable region of the cuff on the medial portion of the thigh covering the femoral artery, it will be progressively inflated, waiting 15 seconds every 30 mmHg until the point at which the auscultatory pulse of the tibial artery is interrupted.

CONTACTS AND LOCATIONS:
Locations (1):
- Franciele Marques Vanderlei, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No